CLINICAL TRIAL: NCT02222480
Title: A 2-Week, Randomized, Double-Blind, Parallel, Placebo-Controlled Study to Evaluate the Efficacy, Tolerability, and Pharmacokinetic-Pharmacodynamic Relationship of Fimasartan in Combination With Hydrochlorothiazide in Patients With Mild to Moderate Hypertension
Brief Title: A Clinical Trial to Evaluate Efficacy, Tolerability, and Pharmacokinetic-Pharmacodynamic Relationship of Fimasartan/Hydrochlorothiazide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Collaborators: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BR-FHC-CT-201-BZ
Record Dates: First submitted 2014-08-18; First posted 2014-08-21 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Hypertension
Keywords: Patients; with mild; moderate; essential
MeSH Terms: conditions — Hypertension; Lymphoma, Follicular | interventions — fimasartan; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Fimasartan 60 mg, Hydrochlorothiazide 12.5 mg (Experimental): Combination of Fimasartan/Hydrochlorothiazide 60/12.5mg
  Interventions: Drug: Fimasartan; Drug: Hydrochlorothiazide
- Fimasartan 60 mg, Hydrochlorothiazide 25 mg (Experimental): Combination of Fimasartan/Hydrochlorothiazide 60/25mg
  Interventions: Drug: Fimasartan; Drug: Hydrochlorothiazide
- Fimasartan 120 mg, Hydrochlorothiazide 12.5 mg (Experimental): Combination of Fimasartan/Hydrochlorothiazide 120/12.5mg
  Interventions: Drug: Fimasartan; Drug: Hydrochlorothiazide
- Fimasartan 120 mg, Hydrochlorothiazide 25 mg (Experimental): Combination of Fimasartan/Hydrochlorothiazide 120/25mg
  Interventions: Drug: Fimasartan; Drug: Hydrochlorothiazide
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fimasartan
  Arms: Fimasartan 120 mg, Hydrochlorothiazide 12.5 mg; Fimasartan 120 mg, Hydrochlorothiazide 25 mg; Fimasartan 60 mg, Hydrochlorothiazide 12.5 mg; Fimasartan 60 mg, Hydrochlorothiazide 25 mg
Drug: Hydrochlorothiazide
  Arms: Fimasartan 120 mg, Hydrochlorothiazide 12.5 mg; Fimasartan 120 mg, Hydrochlorothiazide 25 mg; Fimasartan 60 mg, Hydrochlorothiazide 12.5 mg; Fimasartan 60 mg, Hydrochlorothiazide 25 mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
A 2-Week, Randomized, Double-Blind, Parallel, Placebo-Controlled Study to Evaluate the Efficacy, Tolerability, and Pharmacokinetic-Pharmacodynamic Relationship of Fimasartan in Combination with Hydrochlorothiazide in Patients with Mild to Moderate Hypertension

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects of no childbearing potential 19-70 years of age
2. Mean clinic-measured sitting DBP (siDBP) of 90-109 mmHg and mean clinic-measured sitting SBP (siSBP) of 140-179 mmHg after a ≥1-week washout of prior antihypertensive medications (no wash-out is needed for those not on any antihypertensive medications) with a difference of ≤10 mmHg in sitting DBP between before and after run-in
3. Subjects who agree to participate in this study and give written informed consent
4. Subjects considered to understand the study, be cooperative, and able to be followed-up until the end of the study

Exclusion Criteria:

1. Severe hypertension, i.e., mean siDBP ≥110 mmHg or mean siSBP ≥180 mmHg
2. Orthostatic hypotension with clinically significant signs or symptoms
3. Secondary hypertension
4. Not able to stop administration other antihypertensive medications than the study drugs (i.e., fimasartan and hydrochlorothiazide) throughout the entire study period
5. Clinically significant abnormal laboratory test results, e.g., serum creatinine >1.5 times upper limit of normal, AST, ALT > 2 times upper limit of normal
6. Conditions that may affect to absorption, distribution, metabolism, and excretion for the study drugs
7. Severe insulin-dependent or uncontrolled diabetes mellitus (HbA1c >9%, increased dose of an oral hypoglycemic agent within 12 weeks before screening, or active insulin treatment at screening)
8. Severe cardiovascular diseases within 6 months of screening including ischemic heart disease, peripheral vascular disease, significant ventricular tachycardia, atrial fibrillation, atrial flutter or other significant arrhythmia, hypertrophic obstructive cardiomyopathy, severe obstructive coronary artery disease, aortic stenosis, hemodynamically significant aortic valve or mitral valve disease, severe cerebrovascular disease
9. History of percutaneous transluminal coronary angiography or coronary artery bypass graft
10. Chronic debilitating disease, autoimmune disease, connective tissue disease
11. Positive on serum hepatitis B surface antigen, anti-hepatitis C virus antibody, or anti-HIV antibody
12. History or evidence of alcohol or drug abuse within 2 years
13. Known allergic reaction to any angiotensin receptor blockers
14. Chronic inflammation disease requiring chronic anti-inflammation therapy
15. Women of childbearing potential without any contraceptive measure or breast-feeding mother
16. Prior participation in a clinical trial of any investigational products within 12 weeks from screening
17. Serum potassium <3.5 mmol/L or >5.5 mmol/L at any time of the study period
18. Depletion of sodium ion or body fluid, which cannot be corrected easily during the study period
19. Evidence of hereditary disease, including galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption.
20. Considered unsuitable to participate in the study under the discretion of the principal investigator

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2014-10; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change of treatment in 24-hour mean systolic blood pressure (SBP) using ambulatory blood pressure monitoring (ABPM) | from baseline to 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea